CLINICAL TRIAL: NCT07043751
Title: A Phase I Clinical Trial Evaluating the Tolerance, Pharmacokinetics and Preliminary Efficacy of Injection TQB6411 in Subjects With Advanced Malignant Tumors
Brief Title: A Clinical Trial Evaluating Injection of TQB6411 in Subjects With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB6411-I-01
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-03

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB6411 injection (Experimental): Intravenous injection, the dosage begins on the first day of each cycle, and one treatment cycle every 3 weeks; the dose group is between 0.8 mg/kg-8 mg/kg.
  Interventions: Drug: TQB6411 injection

INTERVENTIONS:
Drug: TQB6411 injection — TQB6411 for injection is an antibody-conjugated drug (ADC) targeting EGFR/c-Met. After injecting intravenously, the antibody part of this product binds to the EGFR and c-Met on the surface of tumor cells to block the activation of EGFR and c-Met signaling pathways. The ADC is enrolled and transported to the lysosome through cells. The linker releases toxins after enzyme cleavage, resulting in DNA damage and cell death.

SUMMARY:
TQB6411 for injection is an antibody-conjugated drug (ADC) targeting EGFR/c-Met. After injecting blood intravenously, the antibody part of this product binds to the surface of EGFR and c-Met on tumor cells to block the activation of EGFR and c-Met signaling pathways. The ADC is enzymatically transported to the lysosome. The linker releases toxins after enzyme cleavage, resulting in DNA damage and cell death. TQB6411 for injection is intended for the treatment of advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed an informed consent form, and had good compliance;
* 18 years old≤age age≤75 years old (calculated based on the date of signing the informed consent form);
* Eastern Cooperative Oncology Group (ECOG) score 0~1 point;
* Expected survival is greater than 12 weeks;
* According to the RECIST v1.1 standard, there is at least one evaluable tumor lesion in the dose escalation stage, and at least one measurable lesion in the dose expansion stage;
* Laboratory examination standards that meet the program requirements (no use of hematopoietic stimulator drugs for correction within 7 days);
* Subjects who failed or were intolerant of standard treatment;
* Subject requirements for the dose expansion stage: advanced NSCLC; metastatic colon cancer; recurrent/metastatic esophageal squamous cell carcinoma; recurrent/metastatic nasopharyngeal carcinoma; advanced malignant solid tumor;
* Can provide tumor tissue specimens that meet the requirements for immunohistochemical testing;
* Women of childbearing age should agree that effective contraception must be adopted during the study period and within 6 months after the end of the study, and that the serum or urine pregnancy test will be negative within 7 days before the study enrollment; men should agree that effective contraception must be adopted within 6 months after the end of the study period;

Exclusion Criteria:

* Have appeared or are currently suffering from other malignant tumors;
* There are diseases that affect intravenous injection and intravenous blood collection;
* The adverse reactions of previous treatments failed to recover to CTCAE V5.0 grade score ≤1, except for toxicity without safety risk, such as grade 2 hair loss, grade 2 peripheral nerve toxicity, grade 2 anemia, non-clinical significance and asymptomatic grade 2 laboratory abnormalities, stable hypothyroidism with hormone replacement therapy;
* Those who have received major surgical treatment, obvious traumatic injury or major surgery during the expected study treatment within 4 weeks before the first medication (except for the surgery stipulated in the program), or have long-term uncured wounds or fractures;
* Subjects with any bleeding or bleeding events ≥CTC AE grade 3 within 4 weeks before the first dose;
* Arterial/venous thrombosis events occurred within 6 months before the first dose;
* People with active viral hepatitis and poor control;
* People infected with active syphilis who need treatment;
* There is a history of active tuberculosis, idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia/radio-pneumonia that needs treatment, or active pneumonia with obvious clinical symptoms, and interstitial lung disease (ILD) that needs treatment, or currently associated with interstitial lung disease;
* Those with a history of abuse of psychotropic substances and cannot quit or have mental disorders;
* Preparing for or having previously received allogeneic bone marrow transplants or solid organ transplants;
* Have a history of hepatic brain disease;
* Suffering from major cardiovascular disease;
* Severe infection that is active or uncontrollable (≥CTC AE grade 2 infection);
* People who require hemodialysis or peritoneal dialysis if renal failure is required;
* Have a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency diseases;
* Subjects who have poorly controlled autoimmune diseases and need to use immunosuppressive agents or systemic hormones to achieve immunosuppressive purposes and still need to continue using them within 7 days before the first dose (except for daily dose of glucocorticoid <10 mg prednisone or other therapeutic hormones);
* People with epilepsy and need treatment;
* Poor diabetes control [fasting blood sugar (FBG) > 10mmol/L];
* Tumor-related symptoms and treatment: subjects who have received chemotherapy, immunotherapy, small molecule targeted drugs, etc. within 3 weeks before the first dose, or are still in the 5 half-life of the drug; within 1 week before the first dose, they have received Chinese patent medicine treatment with anti-tumor indications in the National Medical Products Administration (NMPA) approved drug instructions; imaging (CT or MRI) shows that the tumor has invaded important blood vessels or the researchers judged that the tumor is very likely to invade important blood vessels during the subsequent study and causing fatal major bleeding; if it is not controlled, pleural effusion, pericardial effusion or moderate and severe ascites that still require repeated drainage; known to suffer from spinal cord compression, meningeal metastasis/cancer meningitis, accompanied by brain metastasis symptoms or symptoms/image control time is less than 4 weeks;
* Known allergies to research drugs or excipients;
* Have received previous treatment for Epidermal Growth Factor Receptor (EGFR)/c-Mesenchymal-epithelial transition dual anti-ADC drugs;
* Those who participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first medication;
* According to the researcher's judgment, there are situations that seriously endanger the safety of the subject or affect the subject's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to24 months
  Dosage-limiting toxicity refers to any of the following events that researchers and sponsors believe to be related to the treatment of TQB6411 for injection (including positively related, likely related, and possible related) (except for special instructions, the degree of adverse events is evaluated in accordance with National Cancer Institute (NCI) Common Terminology Criteria (CTC) for Adverse Events (AE) v5.0.
Maximum Tolerated Dose | Up to24 months
  Defined as the highest dose in less than 33% of subjects with dose-limiting toxicity (DLT).
Phase II recommended dose | Up to24 months
  The recommended dose for subsequent phase II studies will be determined based on Maximum Tolerated Dose (MTD), Pharmacokinetics (PK), preliminary efficacy and safety.
Rate and severity of adverse events | Up to24 months
  Rate and severity of adverse events

SECONDARY OUTCOMES:
Peak drug concentration (Cmax) | Within 14 days after administration
  It refers to the highest blood drug concentration achieved after administration of TQB6411 for injection.
Area under the concentration-time curve from time zero to the last measurable concentration time t (AUC0-t) | Within 14 days after administration
  Area under the concentration-time curve from time zero to the last measurable concentration time t (AUC0-t).
Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) | Within 14 days after administration
  Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞).
Peak time (Tmax) | Within 14 days after administration
  It refers to the time when the maximum blood drug concentration is reached after administration of TQB6411 for injection.
Overall response rate (ORR) | Up to 24 months
  Proportion of subjects with best response as Partial relief (PR), Complete Response (CR).
Disease Control Rate (DCR) | Up to 24 months
  Proportion of subjects with best response as Complete Response (CR), Partial relief (PR), Stable Disease (SD).
Progression-free survival (PFS) | Up to 24 months
  The time between the first dose of the trial drug and the date of first definite disease progression or death (from any cause), whichever occurs first.
Overall survival (OS) | Up to 24 months
  Time from first dose of study drug to date of death from any cause.
The incidence of antibiotic-resistant antibodies (ADA) and neutralizing antibodies (NAbs) | Up to 24 months
  The incidence of antibiotic-resistant antibodies (ADA) and neutralizing antibodies (NAbs)

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Dongguan People's Hospital, Dongguan, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangdong, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Anyang Tumor Hospital, Anyang, Henan
  - The Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital Of Wuhan University, Wuhan, Hubei
  - the Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Jining First People's Hospital, Jining, Shandong
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality